CLINICAL TRIAL: NCT00100646
Title: A Randomized Clinical Trial Assessing Continuous HAART Versus Interrupted HAART in a Resource Poor Clinic
Brief Title: Anti-HIV Treatment Interruptions in HIV Infected Adults in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Wistar Institute (Other)
Responsible Party: Principal Investigator, Luis Montaner, Professor and Director, HIV-1 Immunopathogenesis Laboratory, The Wistar Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI051986-01A2 (NIH); R01AI051986 (NIH); Protocol 2411209; 1R01AI051986-01A2 (NIH); R01 A151986-01
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Treatment Interruption; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption; Lamivudine; Lopinavir; Stavudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Highly active antiretroviral therapy (HAART) consisting of lamivudine, lopinavir/ritonovir, and stavudine for 16 weeks with three structured treatment interruptions for 2, 4, and 8 weeks each; rabies vaccine at Weeks 16, 17, 22 and 92.
  Interventions: Behavioral: Structured treatment interruption; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Stavudine; Biological: Rabies de novo antigen
- 2 (Active Comparator): Continuous HAART consisting of lamivudine, lopinavir/ritonovir, and stavudine throughout the study; rabies vaccine at Weeks 16, 17, 22 and 92.
  Interventions: Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Stavudine; Biological: Rabies de novo antigen

INTERVENTIONS:
Behavioral: Structured treatment interruption — Interruptions in treatment will last 2, 4, and 8 weeks in between 16-week periods of ART
  Other Names: STI
  Arms: 1
Drug: Lamivudine — 300 mg tablet taken orally daily
Drug: Lopinavir/Ritonavir — 400 mg lopinavir/100 mg ritonavir tablet taken orally twice daily
Drug: Stavudine — Dosage dependent on weight
Biological: Rabies de novo antigen — Vaccine injected intramuscularly

SUMMARY:
HIV infected people often must take anti-HIV drugs for long periods, leading to long-term drug exposure and toxicity. Interruptions in anti-HIV therapy, also known as structured treatment interruptions (STIs), may have few negative health effects and may be helpful to the overall long-term health of HIV-infected people. The purpose of this study is to determine if sequential short-term STIs of antiretroviral therapy (ART) in HIV infected individuals in a resource-constrained environment can retain the immune reconstitution benefits of continuous treatment while potentially lessening rates of toxicity associated with continuous therapy strategies and at the same time, lessen costs associated with ART.

DETAILED DESCRIPTION:
Long-term toxicity and the high cost of medications are two problems faced by HIV infected people taking ART. Previous studies in HIV-infected patients suggest that ART with STIs may decrease drug exposure and lessen long-term drug toxicity, while not sacrificing viral suppression and patient health. This study will determine if ART with STIs can maintain the same level of immune function in HIV-infected people as continuous ART. This study will recruit patients in South Africa.

This study will last 3.5 years. At study entry, all participants will begin daily ART consisting of lamivudine, lopinavir/ritonavir, and stavudine. At Month 6, only participants who have responded well to ART (CD4 count greater than 450 cells/uL and viral load less than 50 copies/ml at Month 6) will be randomly assigned to one of two groups. Group 1 participants will participate in STIs during therapy, and Group 2 participants will receive continuous therapy. People in Group 1 will have treatment interruptions of 2, 4, and 8 weeks of duration in between 16-week periods of ART. Group 1 participants will re-initiate therapy if their CD4 count drops below 350 cells or evidence of clinical disease progression is present. Group 2 participants will continue taking ART throughout the study.

At screening, participants will undergo medical history assessment, a physical exam, and magnetic resonance imaging (MRI) and dual energy x-ray absorptiometry (DEXA) scans. There will be at least 22 study visits occurring approximately every 8 weeks, each lasting 45 to 60 minutes. At each study visit, participants will be required to bring any remaining pills with them so adherence can be assessed and will undergo medical assessments. Blood collection will occur at nearly all visits. For female participants, urine collection will occur at all visits. Participants will receive rabies vaccinations at Weeks 16, 17, and 22. A visit at Week 92 will include an MRI and participants will receive a rabies vaccine booster.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count of 200 to 350 cells/mm3 within 60 days of starting study treatment
* Antiretroviral naive. Participants who have received antiretrovirals through postexposure prophylaxis or short course therapy to prevent mother-to-child transmission are eligible for this study.
* Willing to adhere to study treatment
* Willing to be followed for the duration of this study

Exclusion Criteria:

* History of AIDS-defining illness (CDC category C). Patients with a history of pulmonary tuberculosis are not excluded.
* Newly diagnosed AIDS-defining opportunistic infection or other condition requiring acute therapy at study entry
* Previous therapy with agents with significant myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic potential within 30 days prior to study entry
* History of immunomodulatory therapy within 4 weeks prior to screening, or cannot abstain from immunomodulators during the study
* Previously received rabies vaccine
* Current alcohol or drug abuse that, in the opinion of the investigator, may interfere with the study
* Diarrhea (more than 6 stools per day for 7 consecutive days) within 30 days prior to study entry
* Active or suspected acute hepatitis within 30 days of study entry
* Bilateral peripheral neuropathy of Grade 2 or higher at screening
* Inability to tolerate oral medication
* Any clinical condition that, in the opinion of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To compare intermittent ART to continuous therapy by comparing endpoint CD4 counts between Groups 1 and 2 | Throughout study
Response to rabies vaccination and booster | Weeks 16, 22, and 92

SECONDARY OUTCOMES:
Comparison of treatment-associated toxicity and safety of 2 to 8 weeks of antiretroviral therapy (ART) interruption versus continuous ART | Throughout study
Determine the outcome of immune reconstitution by monitoring changes in T-cell subsets and the ability to maintain cell-mediated responses against various antigens | Before and after intermittent strategy
Viral evolution and genotypic changes that confer drug resistance | During intermittent and continuous treatment
Effect of treatment interruption on cardiovascular adverse experiences risk factors | From Weeks 0 to 144

CONTACTS AND LOCATIONS:
Overall Officials: Luis J. Montaner, DVM, MSc, DPhil, Principal Investigator — The Wistar Institute; Ian M. Sanne, MBBCH, FCP(SA), DTM&H, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- University of the Witwatersrand, Johannesburg, South Africa

REFERENCES:
- [Background] Arnedo-Valero M, Garcia F, Gil C, Guila T, Fumero E, Castro P, Blanco JL, Miro JM, Pumarola T, Gatell JM. Risk of selecting de novo drug-resistance mutations during structured treatment interruptions in patients with chronic HIV infection. Clin Infect Dis. 2005 Sep 15;41(6):883-90. doi: 10.1086/432881. Epub 2005 Aug 4. PMID 16107990
- [Background] Azzoni L, Papasavvas E, Montaner LJ. Lessons learned from HIV treatment interruption: safety, correlates of immune control, and drug sparing. Curr HIV Res. 2003 Jul;1(3):329-42. doi: 10.2174/1570162033485212. PMID 15046257
- [Background] Kumarasamy N, Flanigan TP, Vallabhaneni S, Cecelia AJ, Christybai P, Balakrishnan P, Yepthomi T, Solomon S, Carpenter CC, Mayer KH. A randomised control trial of structured interrupted generic antiretroviral therapy versus continuous therapy in HIV-infected individuals in Southern India. AIDS Care. 2007 Apr;19(4):507-13. doi: 10.1080/09540120701213849. PMID 17453591
- [Background] Papasavvas E, Grant RM, Sun J, Mackiewicz A, Pistilli M, Gallo C, Kostman JR, Mounzer K, Shull J, Montaner LJ. Lack of persistent drug-resistant mutations evaluated within and between treatment interruptions in chronically HIV-1-infected patients. AIDS. 2003 Nov 7;17(16):2337-43. doi: 10.1097/00002030-200311070-00008. PMID 14571185
- [Background] Papasavvas E, Kostman JR, Mounzer K, Grant RM, Gross R, Gallo C, Azzoni L, Foulkes A, Thiel B, Pistilli M, Mackiewicz A, Shull J, Montaner LJ. Randomized, controlled trial of therapy interruption in chronic HIV-1 infection. PLoS Med. 2004 Dec;1(3):e64. doi: 10.1371/journal.pmed.0010064. Epub 2004 Dec 28. PMID 15630469
- [Result] Azzoni L, Foulkes AS, Firnhaber C, Yin X, Crowther NJ, Glencross D, Lawrie D, Stevens W, Papasavvas E, Sanne I, Montaner LJ. Metabolic and anthropometric parameters contribute to ART-mediated CD4+ T cell recovery in HIV-1-infected individuals: an observational study. J Int AIDS Soc. 2011 Jul 29;14:37. doi: 10.1186/1758-2652-14-37. PMID 21801351
- [Result] Firnhaber C, Azzoni L, Foulkes AS, Gross R, Yin X, Van Amsterdam D, Schulze D, Glencross DK, Stevens W, Hunt G, Morris L, Fox L, Sanne I, Montaner LJ. Randomized trial of time-limited interruptions of protease inhibitor-based antiretroviral therapy (ART) vs. continuous therapy for HIV-1 infection. PLoS One. 2011;6(6):e21450. doi: 10.1371/journal.pone.0021450. Epub 2011 Jun 28. PMID 21738668
- [Result] Foulkes AS, Azzoni L, Li X, Johnson MA, Smith C, Mounzer K, Montaner LJ. Prediction based classification for longitudinal biomarkers. Ann Appl Stat. 2010 Sep;4(3):1476-1497. doi: 10.1214/10-AOAS326. PMID 21274424
- [Result] Azzoni L, Crowther NJ, Firnhaber C, Foulkes AS, Yin X, Glencross D, Gross R, Kaplan MD, Papasavvas E, Schulze D, Stevens W, van der Merwe T, Waisberg R, Sanne I, Montaner LJ. Association between HIV replication and serum leptin levels: an observational study of a cohort of HIV-1-infected South African women. J Int AIDS Soc. 2010 Sep 7;13:33. doi: 10.1186/1758-2652-13-33. PMID 20822522